CLINICAL TRIAL: NCT05692570
Title: A Phase 1, Open-label Drug Interaction Study of PBI-200 With Ritonavir or Cobicistat in Healthy Volunteers
Brief Title: A Study of PBI-200 With Ritonavir or Cobicistat in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pyramid Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBI-200-106
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Drug-drug Interaction
MeSH Terms: interventions — Ritonavir; Cobicistat

STUDY DESIGN:
Intervention Model Description: Single-sequence, three-periods
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single-sequence, 3-period (Experimental): Period 1: single dose of PBI-200; Period 2: daily dosing of ritonavir with a single dose of PBI-200 co-administered once ritonavir steady state reached; Period 3: daily dosing of cobicistat with a single dose of PBI-200 co-administered once cobicistat steady state reached.
  Interventions: Drug: PBI-200 Tablet; Drug: Ritonavir Oral Tablet; Drug: Cobicistat Oral Tablet

INTERVENTIONS:
Drug: PBI-200 Tablet — PBI-200 is a TRK inhibitor
Drug: Ritonavir Oral Tablet — Ritonavir is a potent CYP3A inhibitor
  Other Names: Norvir
Drug: Cobicistat Oral Tablet — Cobicistat is a potent CYP3A inhibitor
  Other Names: Tybost

SUMMARY:
This is a drug-drug interaction study in volunteers to evaluate the effect of ritonavir or cobicistat on the pharmacokinetics (PK) of PBI-200.

DETAILED DESCRIPTION:
This is an open-label, single-sequence, three-period drug-drug interaction study in healthy male and female volunteers to evaluate the effect of a potent CYP3A inhibitor, ritonavir or cobicistat, on the single dose PK of orally administered PBI-200. It is expected that co-administration of ritonavir or cobicistat with PBI-200 will increase the exposure of PBI 200.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 55 years of age (inclusive).
* Body Mass Index (BMI) between 18.0 and 32.0 kg/m² (inclusive).
* Non-smoking/non-vaping, healthy, with no history of clinically relevant medical illness.

Exclusion Criteria:

* History or presence of clinically significant cardiovascular, pulmonary, respiratory, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease which, in the opinion of the Investigator, would jeopardize the safety of the volunteer or impact the validity of the study results.
* History of gastrointestinal/hepatobiliary or other surgery that may affect PK profiles (i.e., hepatectomy, gastric, bypass, or digestive organ resection).
* Intolerance to repeated venipuncture.
* Smoking or use of tobacco products (including vaping) within 3 months prior to the first study drug administration.
* Have a positive drug/alcohol screen, or history or presence of alcoholism or drug abuse within 6 months of first study drug administration.
* Volunteers with a corrected QT using Fridericia's formula (QTcF) prolongation over 450 milliseconds at Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2022-11-12 (Actual); Study Completion 2022-11-12 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration [C(max)] of PBI-200 | 11 days
  Maximum (peak) plasma drug concentration
Area Under the Concentration-Time Curve (AUC) from time zero to the time of the last measurable concentration [AUC(0-t)] | 11 days
  AUC, calculated using linear up / log down trapezoidal method from time zero to time t, where t is the time of the last measurable concentration.
AUC from time zero to infinity [AUC(0-inf)] | 11 days
  AUC from time zero to infinity, AUC(0-inf) = AUC(0-t) + Ct/kel, where kel is the terminal rate constant and Ct is the last measurable concentration.
Terminal elimination half-life [T(1/2)] | 11 days
  Apparent terminal elimination half-life, calculated as ln(2)/kel.
Incidence, frequency and severity of adverse events (AEs) | 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Pyramid Biosciences
Locations (1):
- Celerion, Inc., Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No